CLINICAL TRIAL: NCT07307898
Title: Cavitation Versus Whole-Body Electromyostimulation on Infilamatory Markers in Centeral Obesity
Brief Title: Cavitaion vs W-BEMS on Central Obesity
Acronym: w-bems
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hadeer Elsayed Abdelrazik Elsayed Ramadan, physical therapist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 012/005581
Record Dates: First submitted 2025-08-26; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Central Obesity
MeSH Terms: conditions — Obesity, Abdominal

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group A (Study group) (Experimental): Participants in this cohort were administered localized ultrasound cavitation treatments. Each session was approximately 30 minutes in duration, with treatments scheduled twice a week. In addition, participants received mediterranean diet
  Interventions: Device: cavitation, whole body electromyostimulation
- group B (Study group) (Experimental): : Participants assigned to this cohort underwent whole- body electromyostimulation (WB-EMS) therapy. These sessions were 20 minutes long, also occurring twice weekly. Participants also received mediterranean diet.
  Interventions: Device: cavitation, whole body electromyostimulation
- Group C (Control Group) (Sham Comparator): Participants in this control group receive mediterranean diet. Additionally, they participated in all assessment procedures, ensuring a comprehensive comparative analysis.
  Interventions: Device: cavitation, whole body electromyostimulation

INTERVENTIONS:
Device: cavitation, whole body electromyostimulation — The duration of the study was set for 12 weeks. Assessments were meticulously conducted at both the baseline and the conclusion of the study period to evaluate outcomes across the different groups.

SUMMARY:
The purpose of this study is to compare the effects of ultrasound cavitation and whole-body electromyostimulation (WB-EMS) on inflammatory markers in individuals with central obesity.

DETAILED DESCRIPTION:
Sixty individuals with central obesity were recruited from private clinics. And underwent a screening process to determine their eligibility based on the inclusion and exclusion criteria. Eligible participants were informed about the study details, procedures, potential risks, and benefits before obtaining written informed consent

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-50 years.
* Individuals diagnosed with central obesity, defined as a waist circumference greater than 102 cm in men and 88 cm in women.
* Participants with a stable body weight for at least three months prior to the study.
* No engagement in regular physical activity or weight loss programs in the past six months.
* Willingness to adhere to study protocols and attend all scheduled sessions.

Exclusion Criteria:

* Individuals with chronic diseases other than obesity-related conditions, such as cardiovascular disease, diabetes, or severe hypertension.

  * Pregnant or lactating women.
  * Individuals with implanted electronic devices (e.g., pacemakers).
  * Participants with dermatological conditions or skin infections in the treatment area.
  * Individuals undergoing medication that may affect fat metabolism or inflammatory markers.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-09-05 (Actual); Primary Completion 2024-11-05 (Actual); Study Completion 2026-01-04 (Estimated)

PRIMARY OUTCOMES:
Inflammatory Markers | 3 Monthes
  Measurement of changes in levels of Tumor Necrosis Factor-alpha (TNF-alpha), and Interleukin-6 (IL-6) using ELISA (Enzyme-Linked Immunosorbent Assay) kits.

SECONDARY OUTCOMES:
Waist Circumference | 3 Monthes
  Will be measured at the level of the iliac crest using a standard measuring tape to assess changes in central adiposity.
Body Weight | 3 Monthes
  Standard clinical scales to measure body weight at each visit to track changes over the study period.
Body Mass Index (BMI) | 3 Monthes
  Will be calculated using measured height and weight (kg/m²) to observe changes in overall body mass classification.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Qalyubia Governorate, Egypt